CLINICAL TRIAL: NCT04036760
Title: Implementation and Evaluation of Care Coordination in Linkage to Care for Hepatitis C Following Release From New York City Jails
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 14-02105
Record Dates: First submitted 2019-07-19; First posted 2019-07-30 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard of Care transitional care coordination
- Research transitional care coordination
  Interventions: Behavioral: Research transitional care coordination

INTERVENTIONS:
Behavioral: Research transitional care coordination — Though care coordination was offered to all HCV positive inmates who are approached,the care coordination will still constitute a research intervention that requires informed consent, rather than a new uniform standard of care, to allow maximum autonomy for this incarcerated population.
  Groups: Research transitional care coordination

SUMMARY:
This study assesses the impact of a hepatitis C care coordination program on rates of linkage to hepatitis C care following release from New York City jails. Adult patients (age 18 years and above) with chronic Hepatitis C infection at Bellevue Hospital Center 19 North prison clinic from July 1, 2015 through December 31, 2016 will be offered participation in a transitional care coordination program. The rates of linkage of these individuals following release from jail will be compared to a historical cohort of adult patients with chronic Hepatitis C infection at the 19 North prison clinic from January 1, 2014 through June 31, 2015.

ELIGIBILITY:
Inclusion Criteria:

* HCV infection seen in Bellevue's 19N prison Infectious Diseases clinic.

Exclusion Criteria:

* Individuals who refuse to participate in the study when approached
* Individuals who are unable or unwilling to sign a consent form agreeing to participate. Participants must have sufficient literacy to sign their name, as written informed consent is required for study participation
* Individuals who are unable to successfully negotiate the use of a telephone interpreter if required
* Individuals who have received a sentence that extends beyond the interval of follow up (one year sentence in city jail)
* Individuals who will be moved upstate to prison directly from jail
* Individuals who die prior to discharge from Rikers Island

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males and gender self-identified females age 18 or over with HCV infection seen in Bellevue's 19N prison Infectious Diseases clinic.
Study Population: Males and gender self-identified females age 18 or over with HCV infection seen in Bellevue's 19N prison Infectious Diseases clinic.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
The proportion of adult inmates linked to care following release from jail between the period of January 1st 2014 to January 31st 2014 compared with February 1st 2015 to December 31st 2015 after the implementation of care coordination. | 2 Years

SECONDARY OUTCOMES:
The proportion of those adult inmates who were successfully linked to care at Bellevue Hospital Center (BHC) during the period before and after the implementation of care coordination who subsequently had at least two visits with an HCV provider. | 2 Years
The proportion of those adult inmates who were linked to care at BHC during the period before and after the implementation of care coordination who then initiated Hepatitis C Virus (HCV) treatment. | 2 Years
The proportion of those adult inmates who were linked to care at BHC during the period before and after the implementation of care coordination who then went onto achieve an Sustained Virologic Response (SVR) when treated. | 2 Years
The proportion of those adult inmates who were linked to care at BHC during the period before and after the implementation of care coordination who were linked to ancillary services. | 2 Years
Retention in care as defined as two sequential clinic ID clinic visits during 12 months | 2 Years
  Number of patients who are able to retain 2 sequential visits during 12 months
Documented sustained virologic response (SVR) | 2 Years
  no detectable RNA in 2 years post treatment
Documented sustained HCV cure | 2 Years
  Showing no symptoms of HCV for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Eckhardt, MD, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

REFERENCES:
- [Derived] Akiyama MJ, Columbus D, MacDonald R, Jordan AO, Schwartz J, Litwin AH, Eckhardt B, Carmody E. Linkage to hepatitis C care after incarceration in jail: a prospective, single arm clinical trial. BMC Infect Dis. 2019 Aug 8;19(1):703. doi: 10.1186/s12879-019-4344-1. PMID 31395019